CLINICAL TRIAL: NCT03690453
Title: Open-Label Study to Evaluate Pharmacokinetic Properties and Mosquito-Lethal Effect of Ivermectin Metabolites in Healthy Adult Subjects
Brief Title: Effect of Ivermectin Metabolites on Mosquito Survival
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MAL18006
Record Dates: First submitted 2018-09-18; First posted 2018-10-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteer for Clinical Trial (Experimental)
  Interventions: Drug: Ivermectin
- Healthy volunteer for blood donor (No Intervention)

INTERVENTIONS:
Drug: Ivermectin — single dose of Ivermectin
  Arms: Healthy volunteer for Clinical Trial

SUMMARY:
This clinical trial will be designed to capture the full duration of mosquito-lethal effect of single dose Ivermectin to aid efforts to characterize metabolites with mosquito-lethal effect. Ivermectin and its metabolites likely have antiparasitic properties against asexual and sexual stage Plasmodium parasites that will be investigated with plasma samples from this study.

This is an open-label pharmacokinetic study. Ten healthy participants will be admitted in the inpatient ward to receive a single oral dose of IVM (400 µg/kg).

Another 10 healthy participants will be donate blood up to 42 ml each times for up to 3 times. There is no drug administration for these participants.

The total duration for each volunteer's participation in the study is approximately 2 months.

DETAILED DESCRIPTION:
HEALTHY PARTICIPANT FOR CLINICAL TRIAL

Study will enroll 10 Thai healthy participants, 5 male and 5 female, aged 18-60 years.

Participants will be admitted in the inpatient ward to receive a single oral dose of IVM (400 µg/kg).

After a volunteert has provided written informed consent, the investigator will determine if the volunteer is eligible for enrollment in the study. This will be done by reviewing the inclusion and exclusion criteria and completing all of the screening assessments. Screening assessments may be carried out over more than one day, provided that all required assessments are completed within the 14 days prior to admission for Ivermectin administration.

The blood collection for Standard Membrane Feeding Assay, Direct Feeding Assays, Pharmacokinetic analysis, Plasma for Plasmodium assays and mosquito IgG assays should be obtained at the scheduled times relative to when the participant was dosed.

The total duration for each volunteer's participation in the study is approximately 2 months.

HEALTHY PARTICIPANT FOR BLOOD DONOR

Study will enroll 10 healthy participants, aged 18-60 years. Each participant will donate blood up to 42 ml via venipuncture up to three blood donations. There will be at least 28 days between each blood donation from the same subject.

Blood will be maintained at 37°C in a warm water bath until mixed with ivermectin compounds or metabolites by Pharmacology staff and fed to mosquitoes by Armed Forces Research Institute of Medical Sciences (AFRIMS) staff. Any remaining blood after SMFAs will be discarded. No blood samples will be transferred to AFRIMS. Participants for blood donation should not be the same participants enrolled in the clinical trial above.

ELIGIBILITY:
Inclusion Criteria for Ivermectin intervention group:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females aged between 18 years to 60 years.
3. Males and Females weight between 36-75 kilograms.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Provide a signed and dated written informed consent prior to study participation.
7. Willingness and ability to comply with the study protocol for the duration of the trial.
8. Able to tolerate direct mosquito feeding.
9. Blood hemoglobin in males >13 g/dL and females >12 g/dL.
10. Normal electrocardiogram (ECG) with QTc <450 msec.

Exclusion Criteria for Ivermectin intervention group:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. A positive hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
3. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes (heart failure, hypokalemia) or with a family history of sudden cardiac death.
4. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   Clcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
5. History of alcohol or substance abuse or dependence within 6 months of the study.
6. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions
7. Use of prescription (especially CYP3A4 inhibitors or inducers) or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins (especially vitamin C), herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Plasma donation during the study is not acceptable.
11. Subjects who have a history of allergy to IVM, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. AST or ALT >1.5 upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. History of IVM or other drug treatments known to be CYP3A4 inducers or inhibitors (e.g. piperaquine, ritonavir, rifampicin) within 3 months.
16. The subject is unwilling to abstain from the consumption of food containing vitamin C (e.g. fruits, juices, papaya salad) 12 hours before and after drug ingestion.
17. History of travel to West or Central Africa, unless it can be verified that subject does not have Loa loa infection.
18. History or suspected of hypersensitivity/anaphylaxis to mosquito bites and other insect bites/sting (e.g. history of cellulitis-like cutaneous inflammation, anaphylaxis, hives)

Inclusion criteria for healthy blood donor:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females aged between 18 years to 60 years.
3. Males and Females weight between 36-75 kilograms.
4. Provide a signed and dated written informed consent prior to study participation.
5. Willingness and ability to donate blood.

Exclusion criteria for healthy blood donor:

1. Females who are pregnant, trying to get pregnant, or are lactating (determined by verbally asking and urine pregnancy test).
2. The subject has evidence of active substance abuse that may compromise safety or ability to adhere with protocol instructions.
3. A positive hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. History of alcohol or substance abuse or dependence within 6 months of the study.
5. Any known blood disorders (e.g. thalassemia, sickle cell anemia)
6. Use of prescription (especially CYP3A4 inhibitors or inducers) or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins (especially vitamin C), herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to blood collection unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
7. The subject has participated in a clinical trial and has received a drug (particularly IVM or any drug known to be a CYP3A4 inducer or inhibitor) or a new chemical entity within 90 days prior to blood collection.
8. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to blood collection.
9. The subject is unwilling to abstain from consumption of food containing vitamin C (e.g. fruits, juices, papaya salad within 12 hours prior to blood collection.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve for Ivermectin and its metabolites | 41 days
  Pharmacokinetic parameters (area under the concentration-time curve [(AUC∞ and AUCLAST] for Ivermectin and its metabolites.
Maximum concentration for Ivermectin and its metabolites | 41 days
  Pharmacokinetic parameters (maximum concentration [CMAX]) for Ivermectin and its metabolites.
Time to maximum concentration for Ivermectin and its metabolites | 41 days
  Pharmacokinetic parameters (time to maximum concentration [TMAX]) for Ivermectin and its metabolites.
Terminal elimination half-life for Ivermectin and its metabolites | 41 days
  Pharmacokinetic parameters (terminal elimination half-life [t1/2]) for Ivermectin and its metabolites.
Concentration associated with half maximum mosquito killing effect [LC50] for Ivermectin and its metabolites | 41 days
  Pharmacodynamic parameters (concentration associated with half maximum mosquito killing effect [LC50]) for Ivermectin and its metabolites.

SECONDARY OUTCOMES:
Duration of mosquito survivorship | 14 days
  Duration of mosquito survivorship following standard membrane feeding assay (SMFA) to determine duration of time post drug administration that IVM-treated volunteers are lethal to An. dirus and An. minimus.
Compare Maximum Blood Concentrations (Cmax) for ivermectin components and metabolites measured between venous and capillary blood | 41 days
  Pharmacokinetic differences for Ivermectin and metabolites in venous and capillary blood.
Compare Area-Under-Curve (AUC) for ivermectin components and metabolites measured between venous and capillary blood | 41 days
  Pharmacokinetic differences for Ivermectin and metabolites in venous and capillary blood.
Compare mosquito (An. dirus) survival curves to day 14 between Direct Feeding Assay and Standard Membrane Feeding Assays | 14 days
  Mosquito survival curves to day 14 within a species will be compared between mosquitoes blood fed via Direct Feeding Assay and Standard Membrane Feeding Assays by Log-Rank survival curve analysis (Mantel-Cox method). This will assess if venous blood is more or less lethal to mosquitoes than blood ingested from subdermal capillaries.
Compare mosquito (An. Minimus) survival curves to day 14 between Direct Feeding Assay and Standard Membrane Feeding Assays | 14 days
  Mosquito survival curves to day 14 within a species will be compared between mosquitoes blood fed via Direct Feeding Assay and Standard Membrane Feeding Assays by Log-Rank survival curve analysis (Mantel-Cox method). This will assess if venous blood is more or less lethal to mosquitoes than blood ingested from subdermal capillaries.
The lethal concentration that kills 50% of mosquitoes (LC50) between two strains of An. dirus | 14 days
  The lethal concentration that kills 50% of mosquitoes (LC50) between two strains of An. dirus will be evaluated. This will assess if one An. dirus strain is more or less susceptible to ivermectin.
Mosquito survival curves to day 14 between two strains of An. dirus. | 14 days
  Mosquito survival curves to day 14 between two strains of An. dirus will be evaluated. This will assess if one An. dirus strain is more or less susceptible to ivermectin.
The lethal concentration that kills 50% of mosquitoes (LC50) for each ivermectin component and synthesized metabolites | 14 days
  The lethal concentration that kills 50% of mosquitoes (LC50) for each ivermectin component and synthesized metabolites. The LC50s and their corresponding 95% confidence intervals will be evaluated for each ivermectin component and synthesized metabolites. This will assess if any of the ivermectin components or metabolites are more or less lethal to An. dirus.
The inhibitory concentration that kills 50% of parasites (IC50) for each P. falciparum strain. | 48 hours
  The inhibitory concentration that kills 50% of parasites (IC50) will be evaluated for each P. falciparum strain to determine which strains are more or less susceptible to ivermectin.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With subject's consent, subject's data and results from blood analyses stored in the database may be shared with other researchers to use in the future.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Kobylinski KC, Tipthara P, Wamaket N, Chainarin S, Kullasakboonsri R, Sriwichai P, Phasomkusolsil S, Hanboonkunupakarn B, Jittamala P, Gemmell R, Boyle J, Wrigley S, Steele J, White NJ, Tarning J. Author Correction: Ivermectin metabolites reduce Anopheles survival. Sci Rep. 2024 Oct 24;14(1):25243. doi: 10.1038/s41598-024-76902-z. No abstract available. PMID 39448768